CLINICAL TRIAL: NCT02076984
Title: LAPAROSCOPIC VENTRAL HERNIA REPAIR BY LIGHTWEIGHT POLYPROPYLENE MESH. A PROSPECTIVE ITALIAN MULTICENTRIC RANDOMIZED STUDY COMPARING TWO FIXATION DEVICES: TITANIUM SPIRAL TACKS vs ABSORBABLE TACKS
Brief Title: Titanium vs Absorbable Tacks for Mesh Fixation in Laparoscopic Incisional and Ventral Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, Gianfranco Silecchia, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11041974
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Ventral Hernia; Incisional Hernia
Keywords: Ventral hernia; Incisional hernia; Patient affected by ventral or incisional hernias
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): laparoscopic incisional or ventral hernia repair use of lightweight polypropylene mesh fixed by titanium tacks
  Interventions: Procedure: Laparoscopic incisional or ventral hernia repair
- Group B (Other): laparoscopic incisional or ventral hernia repair use of lightweight polypropylene mesh fixed by U shaped absorbable tacks
  Interventions: Procedure: Laparoscopic incisional or ventral hernia repair

INTERVENTIONS:
Procedure: Laparoscopic incisional or ventral hernia repair

SUMMARY:
Background: Laparoscopic repair of ventral hernias has gained popularity, since many studies and a recent meta-analysis have reported encouraging results and recurrence rates similar to open repair. The choice of the mesh and fixation methods is of paramount importance during laparoscopic approach, and nowadays, lightweight macropore meshes specifically designed for laparoscopic approach represent the first choice in several studies, due to the biomechanical properties and the optimal integration into the abdominal wall. No data with statistical relevance exist on the choice of fixation methods.

Primary end point of the present Italian multicentric prospective randomized trial is to evaluate the safety and effectiveness of two different tacks to fix the lightweight polypropylene mesh (Physiomesh™) during laparoscopic incisional hernia repair: metallic spiral tacks (Protack™) vs absorbable "U" shaped tacks (Securestrap™)

Design of the Study: 200 patients with ventral hernia will be randomized into two groups:

Group A patients will be submitted to laparoscopic repair by Physiomesh fixed by Protack; Group B patients will be submitted to laparoscopic repair by Physiomesh fixed by Securestrap.

Blind randomization will be guaranteed by an on-line software with specific key access for every surgical unit participating in the study. Patients demographics and characteristics, preoperative studies, intraoperative and postoperative results and complications, as well as scheduled follow-up will be recorded and uploaded to the database. Data represented by continuous variables will be expressed as arithmetic mean +/- standard deviation. Other data will be expressed as geometric mean +/- 95% confidence interval. Data representing low incidence events will be expressed as number and percentage of occurrence for each group. Statistical significance for all analyses will be indicated by a p value of 0.05 or less.

DETAILED DESCRIPTION:
BACKGROUND During the past 50 years, incisional and ventral hernia repair surgery has evolved from direct suture repair to the use of synthetic mesh in order to obtain a tension-free repair (1-3). Finally the tension-free concepts have been applied to laparoscopic surgery. Laparoscopic repair of ventra/incisional hernias has gained increasing popularity, since many studies and a recent meta-analysis and consensus conferences have reported encouraging results, in terms of wound infection, hospital stay and post-operative pain with recurrence rate comparable with open approach (1-7).

Patient selection (age, sex, comorbidities, obesity, hernia site and size, eventual recurrence and type of previous abdominal surgery), choice of the mesh (bio-materials, size and shape) and fixation methods (titanium tacks, absorbable tacks, fibrin glue) are considered crucial issues in preventing recurrence and complications as well as patients compliance and acceptance (4-5, 8-9). The choice of the mesh to implant is of paramount importance, in open as well as in laparoscopic approaches. During the last decade, many meshes and fixation devices have been proposed and tested as a tool to enhance primary and incisional/ventral hernias repair (10-11). Light-weight meshes have been proposed in order to reduce the mesh and/or mesh fixation related complications (12). Decreasing the density of non-absorbable material a reduced "foreign-body response" has been postulated, resulting in improved abdominal wall compliance, less mess shrinkage, thus allowing a better integration in host tissues (13-14).

The "lightweight approach" is also based on the results of studies concerning the abdominal wall biomechanics (15-16) suggesting the characteristics of the "ideal mesh" (elasticity, tensile strength and pressure resistance) similar to the normal abdominal wall. The ideal mesh, should be elastic enough to comply with the movements and elongation of the different areas of the abdominal wall, yet rigid enough to avoid the herniation of the mesh itself, and strong to resist in its position, without degradation, deformation (shrinkage) or creation of defects, life-long.

Among the great amount of meshes and materials utilized for laparoscopic repair, macropore lightweight polypropylene has been demonstrated to be more efficient than other materials (including heavy weight polypropylene) in terms of inflammatory response and mesh integration on host tissues (17-21). The other crucial issue inlaparoscopic repair is the choice of the mesh fixation method: the most commonly used include metal spiral tacks set in a double crown configuration (22-26). Absorbable tacks have been recently introduced (27) in order to improve biocompatibility, reduce the risk of endoperitoneal adhesions due to the presence of metallic tacks, and reduce mid- and long-term postoperative pain. The rationale of the use of absorbable tacks in laparoscopic incisional/ventral hernia repairusing lightweight macropore polypropylene meshes is in the biochemical and biomechanical mesh features, since these meshes become well integrated into the abdominal wall and do not need permanent fixation devices. To date, only two retrospective studies dealing with the clinical use of absorbable tacks with lightweight macropore polypropylene mesh have been published (28-29). The authors report similar results comparing absorbable vs non absorbable tacks in terms of intraoperative and early post-operative results (29). These studies have the pitfalls to be retrospective evaluation on a small series of patients, so the reported results still need to be validated by larger series and prospective study.

THE PRIMARY END POINTS of this prospective multicentric randomized study are:

* compare mid and long-term results of the use of metallic tacks and absorbable tacks to fix lightweight polypropylene mesh during laparoscopic incisional/ventral hernia repair, in terms of hernia recurrence, in order to establish the safety and effectiveness of absorbable tacks;
* compare intraoperative and early port-operative outcomes, in terms of surgical complications, post-operative stay, return to normal life activities and pain management.

METHODS/STUDY DESIGN The prospective randomized multicentric trial will involve 6 Surgical Unit having large experience in laparoscopic incisional/ventral hernia repair and in the use of lightweight polypropylene meshes and both metallic and absorbable tacks (out of the learning curve).

The Referral Centre (General Surgery Unit, ICOT Hospital, Latina, Italy), will coordinate the study and will be responsible of the data analysys and interim evaluation (12 months).

200 patients will be included in the study (see inclusion criteria on table 1), divided into two groups based on an real-time randomization:

* Group A: patients candidate to laparoscopic incisional/ventral hernia repair by lightweight polypropylrne mesh fixed by metallic tacks;
* Group B: patients candidate to laparoscopic incisional/ventral hernia repair by lightweight polypropylene mesh fixed by absorbable tacks.

Blind Randomization will be guaranteed by a dedicated website having restricted access by a password for each surgical unit participating in the study.

All patients will be evaluated by clinical examination, and abdominal CT scan or US scan, in order to evaluate size and number of the defect(s).

All devices used in the study (meshes and tacks) will be:

* Physiomesh™ (Ethicon Endo-Surgery, Johnson & Johnson, Inc) a lightweight polypropylene mesh with double face absorbable layer made to be placed on the peritoneal surface and prevent adhesions with visceral structures;
* Protack™ (Covidien surgical, Mansfield MA, USA), permanent titanium spiral tacks;
* Securestrap™ (Ethicon Endo-Surgery, Johnson & Johnson, Inc), "U"-shaped absorbable tacks made by polydioxanone, which are completely absorbed within 12-18 months after implant.

All procedures will be carried out using the same surgical technique to implant and fix the mesh (overlapping the defect for at least 3 cm on each side), with the tacks set in a double crown configuration at the distance of 1,5 cm , no use of transfixed sutures or glue. After surgery, compressive dressing will be placed for 4 weeks.

A record form (included at the bottom) will be filled for each patient, and sent to the coordinating centre after the patient discharge.

Follow up schedule:

* 1 week (clinical evaluation)
* 4 weeks (clinical evaluation at dressing removal)
* 6 months (clinical evaluation or phone interview)
* 12 months (phone call and eventual clinical evaluation)
* 24 months after surgery (phone call and eventual clinical evaluation)
* 36 months after surgery (phone call and eventual clinical evaluation)

The following parameters will be evaluated:

* Patients characteristics (sex, age, comorbidities, personal therapy)
* Hernia features (location and size)
* Mesh size
* Type of tacks
* Number of tacks
* Operating time
* Post-operative course
* Post-operative complications (according to Clavien-Dindo classification)
* Acute Post-operative pain (using the Visual Numeric Scale for pain classification)
* Return to life activities
* Recurrence rates
* Chronic pain

Data represented by continuous variables (Age, operating time, etc.) will be expressed as arithmetic mean +/- standard deviation. Because of its skewed nature, other data, such as length of hospital stay, pain evaluated by Visual Numeric Scale, will be expressed as geometric mean +/- 95% confidence interval (CI). Other data, such as wound infection, hernia recurrence and other events having low incidence, will be expressed as number and percentage of occurrence for each group.

Statistical significance for all analyses will be indicated by a p value of 0.05 or less. Analysis will be performed by a dedicated software (SAS latest release for Windows).

Table 1: Inclusion criteria

Hernia site* M2 M3 M4 L2 L3 Hernia width* W1 W2 No previous vnetral/incisional hernia repair (R0)* No incarcerated/strangulated hernia No contaminated field or bowel resection during repair BMI < 35 Age between 18 and 75 years old No severe COPD No autoimmune disease under corticosteroids treatment No cirrhosis Child B or C No uncontrolled diabetic (Glycated Hemoglobin < 7)

*: According to: Muysoms FE, et al. Classification of primary and incisional abdominal wall hernias: Hernia 2009; 13: 407-414

ELIGIBILITY:
Inclusion Criteria:

Table 1: Inclusion criteria Hernia site*

* M2
* M3
* M4
* L2
* L3 Hernia width*
* W1
* W2
* No previous vnetral/incisional hernia repair (R0)*
* No incarcerated/strangulated hernia
* No contaminated field or bowel resection during repair
* BMI < 35
* Age between 18 and 75 years old
* No severe COPD
* No autoimmune disease under corticosteroids treatment
* No cirrhosis Child B or C
* No uncontrolled diabetic (Glycated Hemoglobin < 7)

  * According to: Muysoms FE, et al. Classification of primary and incisional abdominal wall hernias: Hernia 2009; 13: 407-414

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
compare mid and long term results in terms of hernia recurrence | 3 years after surgery
  The primary outcome measure will be to assess the incidence of hernia recurrence in both study groups

SECONDARY OUTCOMES:
The secondary outcome measure will be the post-operative pain management | 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medico-Surgical Sciences and Biotechnologies, Sapienza University of Rome, Latina, Italy

REFERENCES:
- [Background] Cavallaro G, Campanile FC, Rizzello M, Greco F, Iorio O, Iossa A, Silecchia G. Lightweight polypropylene mesh fixation in laparoscopic incisional hernia repair. Minim Invasive Ther Allied Technol. 2013 Sep;22(5):283-7. doi: 10.3109/13645706.2013.808228. Epub 2013 Jun 30. PMID 23808370
- [Derived] Silecchia G, Cavallaro G, Raparelli L, Olmi S, Baldazzi G, Campanile FC. Titanium versus absorbable tacks comparative study (TACS): a multicenter, non-inferiority prospective evaluation during laparoscopic repair of ventral and incisional hernia: study protocol for randomized controlled trial. Trials. 2015 Jun 4;16:249. doi: 10.1186/s13063-015-0779-x. PMID 26037907